CLINICAL TRIAL: NCT00171756
Title: A Double-blind, Double-dummy, Multi-centre, Randomized, Active Controlled, Parallel Group Pilot Trial to Compare the Effects of Valsartan and Atenolol on the Pro-thrombotic State in Patients With Mild to Moderate Hypertension.
Brief Title: Study to Compare the Effect of Valsartan vs Atenolol on Pro-thrombotic State in Hypertensive Patients.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CVAL489AGB09
Record Dates: First submitted 2005-09-13; First posted 2005-09-15 (Estimated); Last update posted 2017-02-23 (Actual); Status verified 2017-02

CONDITIONS: Hypertension
Keywords: hypertension; valsartan
MeSH Terms: conditions — Hypertension | interventions — Valsartan; Atenolol

INTERVENTIONS:
Drug: valsartan/atenolol

SUMMARY:
A study to compare the effects of Diovan or Atenolol taken for 12 weeks on platelet function of patients who have mild to moderately severe hypertension

ELIGIBILITY:
Inclusion Criteria:

* Male or female, aged between 18 - 75 years of age inclusively.
* Mild to moderate hypertension (MSDBP >= 95 and >= 110 mmHg and / or MSSBP >140mm Hg) at visit 1, requiring pharmacological intervention. For newly diagnosed patients, hypertensive blood pressure values must be noted on at least two successive examinations prior to entry into the study. In addition, patients must require therapy despite having been following dietary & lifestyle advice for at least 3 months.
* Written informed consent to participate in the study, prior to any study procedures.
* Ability to communicate and comply with all study requirements

Exclusion Criteria:

* o Uncontrolled hypertension defined as seated blood pressure of either systolic BP >180 mmHg and/or diastolic BP >110mmHg.

  * Clinically significant laboratory abnormalities that may interfere with the assessment of safety and/or efficacy of the study drug
  * Patients with severe medical condition(s) that in the view of the investigator may prohibit participation in the study
  * Renal artery stenosis
  * Diabetes Mellitus
  * Any condition resulting from or leading to platelet or clotting abnormalities (eg. hemophilia, von Willebrand's disease).
  * History of a vascular event or intervention (e.g. MI, PTCA or CABG) within 6 months preceding the study.
  * History of clinically significant angina, LVH, transient ischemic attack, stroke, intermittent claudication, deep vein thrombosis (DVT), pulmonary embolism or peripheral vascular disease.
  * Uncontrolled atrial fibrillation (>100 b.p.m. at rest) or other conditions which may require anti-aggregant or anti-vitamin K therapies.
  * Clinical evidence of congestive heart failure.
  * Evidence of second or third degree heart block or sick sinus syndrome.

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2004-06; Primary Completion 2006-03 (Actual); Study Completion 2006-03 (Actual)

PRIMARY OUTCOMES:
Change from baseline in a clinical laboratory measurement of a blood clotting factor after 12 weeks

SECONDARY OUTCOMES:
Change from baseline in clinical laboratory measurements of blood clotting factors, including platelet activation, thrombosis, fibrinolysis, anticoagulation after 12 weeks
Blood pressure of 140/85 mmHg or lower after 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Novartis, Study Director — Novartis
Locations (1):
- Novartis, Basel, Switzerland